CLINICAL TRIAL: NCT00154661
Title: Evaluation of Clinical Efficacy of Pentoxifylline on Patients With Glomerulonephritis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 152S2
Record Dates: First submitted 2005-09-08; First posted 2005-09-12 (Estimated); Last update posted 2005-09-12 (Estimated); Status verified 2001-06

CONDITIONS: Primary Glomerulonephritis
Keywords: glomerulonephritis
MeSH Terms: conditions — Glomerulonephritis | interventions — Pentoxifylline

INTERVENTIONS:
Drug: pentoxifylline

SUMMARY:
we hypothesize that PTX might be effective in lowering proteinuria by modulating renal MCP-1 production in human glomerulonephritis.

DETAILED DESCRIPTION:
Pentoxifylline (PTX) is a phosphodiesterase inhibitor that is widely used for the treatment of peripheral vascular occlusive disorders. In addition, PTX has shown its ability to attenuate nephrotic syndrome secondary to membranous glomerulonephritis and lupus nephritis, and to reduce subnephrotic proteinuria due to early and advanced diabetic nephropathy. However, data with respect to its effect on non-nephrotic primary glomerular diseases are lacking. Moreover, while the anti-proteinuric effect of PTX has been largely attributed to down-regulation of TNF-a, it remains unknown whether other mediators, especially MCP-1, are also affected by PTX. Because our previous works have shown that PTX attenuates proteinuria and suppresses renal MCP-1 mRNA expression in experimental glomerulonephritis in rats, we hypothesize that PTX might be effective in lowering proteinuria by modulating renal MCP-1 production in human glomerulonephritis. This study was thereby conducted to investigate the potential anti-proteinuric and anti-MCP-1 effects of PTX in subnephrotic patients with primary glomerular diseases.

ELIGIBILITY:
Inclusion Criteria:

* glomerular diseases with subnephrotic proteinuria

Exclusion Criteria:

* DM, hepatitis, systemic immunologic renal diseases

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20
Dates: Start 2000-01; Study Completion 2001-06

PRIMARY OUTCOMES:
proteinuria

SECONDARY OUTCOMES:
inflammatory mediators

CONTACTS AND LOCATIONS:
Overall Officials: Pan-Chyr Yang, Study Chair — Professor and vice-Dean
Locations (1):
- Yung-Ming Chen, Taipei, Taiwan